CLINICAL TRIAL: NCT02071654
Title: Efficacy and Safety Evaluation of Transcatheter Pulmonary Valve Implantation for Right Ventricular Outflow Tract (RVOT) Stenosis After Congenital Heart Defect Surgical Correction Complicated With Severe Pulmonary Regurgitation
Brief Title: Efficacy and Safety of Venus P-valve to Treat RVOT Stenosis With Pulmonary Regurgitation
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Venus MedTech (HangZhou) Inc. (Industry)
Collaborators: Core Medical (Beijing) Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VEN2013-10/V2.0
Record Dates: First submitted 2014-01-11; First posted 2014-02-26 (Estimated); Last update posted 2015-01-06 (Estimated); Status verified 2015-01

CONDITIONS: Right Ventricular Outflow Tract Stenosis
Keywords: Venus P-valve

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Venus P-valve transcatheter implantation (Experimental): Single arm of percutaneous implantation of Venus-P valve for treating RVOT stenosis
  Interventions: Device: Venus P-valve transcatheter implantation

INTERVENTIONS:
Device: Venus P-valve transcatheter implantation — Percutaneous implantation of Venus-P valve to treat RVOT stenosis patients

SUMMARY:
A prospective, non-randomized, multi-center clinical study of the Venus P-valve for the treatment of RVOT stenosis with pulmonary regurgitation after surgery of congenital heart defect.

DETAILED DESCRIPTION:
The aim of this protocol is to assess the efficacy, safety and performance of Venus P-valve.

Patients between 18-60 years with RVOT stenosis and moderate to severe pulmonary regurgitation (≥3+) who have undergone trans-annular patch repair of their RVOT, cardiac magnetic resonance (CMR) screening right ventricular end-diastolic volume index (RVEDVI) between 130-160mL/m2.

Post-procedure follow-ups will be scheduled at 24 hours, 30 days, 6 months and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* RVOT stenosis who have undergone transannular patch repair with moderate to severe pulmonary regurgitation
* Isotopic or CMR criteria of RVEDVI≥130mL/m2 and ≤160mL/m2
* Age≥18 years and ≤60 years (Zhongshan Hospital age≥18 years and ≤60 years
* Body weight≥18 kg
* Pulmonary annular diameter between 14mm to 31mm
* RVOT length≥20mm
* The subject or his/her legal representative has provided written informed consent
* Subject will comply with protocol required follow-ups

Add any of the following conditions:

* Subject is symptomatic
* Subject presents with >30% pulmonary regurgitation fraction as defined by cardiac MRI
* ≥3+ pulmonary regurgitation by echocardiograms
* Deteriorating RVEF%
* Progressive tricuspid valve regurgitation (at least moderate degree)
* Complicated with RVOT obstruction (RV systolic pressure>80mmHg)
* Persistent arrhythmias

Exclusion Criteria:

Candidates will be excluded from the study if any of the following conditions are present:

* Existing pulmonary artery branch stenosis or artificial pulmonary valve
* Severe chest wall deformity
* ADHF
* Active infection or endocarditis requiring antibiotic therapy
* Leukopenia (WBC<3000mm3)
* Acute or chronic anemia (Hb<9g/L)
* Platelet account <100,000 cells/mm3
* In the judgment of the investigator, percutaneous introduction and delivery of the valve is not feasible
* A known hypersensitivity to aspirin or heparin
* Positive urine or serum pregnancy test in female subjects
* Ileofemoral vessel characteristics that would preclude safe placement of introducer sheath

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 44 (Estimated)
Dates: Start 2014-02; Primary Completion 2015-02 (Estimated); Study Completion 2016-02 (Estimated)

PRIMARY OUTCOMES:
Improvement rate of RVEDV at 6 months post-procedure. | At 6 months post-implantation of Venus-P valve
  The improvement is defined as the RVEDVI≤108mL/m2 measured with CMR.

SECONDARY OUTCOMES:
Safety Endpoints | From the date of implantation until 12 months post-procedure
  Accumulated occurrences (rate of patients/year) of procedure-related clinical events (death, severe arrhythmias, cardiac tamponade, RVOT or pulmonary artery perforation or rupture, cardiac shock, endocarditis from the date of valve implantation up to 12 months post-procedure or bleeding due to use of heparin/aspirin at 48 hours post-procedure assessed per protocol.
  Occurrence of all deaths (cardiac death, non-cardiac deaths and other deaths) and stroke one year post-procedure.

OTHER OUTCOMES:
Feasibility and Performance Endpoints | Day 7 post-implantation
  Immediate success of implantation of the device measured in percentage (placement of the device and functional stability measured with angiography and hemodynamic performance).
  Function normal of the P valve measured in percentage without major adverse events at day 7.
  (Function normal defined as the P valve's position and function are normal through exams of electrocardiography (EKG), transthoracic echocardiogram (TTE), chest X-ray. )
Secondary Endpoints | From the date of valve implantation till 12 months post-procedure
  Changes of images and clinical parameters pre- and post-procedure at 12 months.
  * CMR: right ventricular volume (expressed as ml/m2), RV ejection fraction (expressed as percentage), pulmonary regurgitation (functional classification as grade I, IIa, IIb and III).
  * Echo: device position(expressed as percentage), hemodynamic performance of velocity of RVOT and pulmonary valve (expressed as m/s), transvalvular pressure gradient, peak pulmonary valve gradient, mean gradient (expressed as the difference of pressure in mmHg.)
  * NYHA class

CONTACTS AND LOCATIONS:
Overall Officials: Junbo Ge, Prof., MD., Principal Investigator — Fudan University
Locations (1):
- Zhongshan Hospital Fudan University, Shanghai, Shanghai Municipality, China